CLINICAL TRIAL: NCT06415175
Title: Prospective, Observational, Longitudinal Study in Paediatric Patients With AD, Treated With Dupilumab in Spain
Brief Title: Study in Paediatric Patients With Atopic Dermatitis Treated With Dupilumab in Spain
Acronym: PROADAP
Status: Recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS18427; U1111-1306-7579 (Registry Identifier: ICTRP)
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Atopic Dermatitis
Keywords: Pediatric
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dupilumab: The information will be collected during consultation as part of the patient's usual follow-up.
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — This study will not administer any treatment, only observe the treatment as prescribed in real world-clinical practice.

SUMMARY:
This is a multicentre, prospective, non-interventional study that aims to describe the treatment patterns of in Atopic dermatitis (AD) patients aged 6 months to 11 years old in Spain: patients' characteristics, disease characteristics, prior treatments for and treatment prescription modalities. As well as to document the real-world effectiveness and safety of dupilumab during the two years of follow up. No diagnostic or therapeutic intervention outside of routine clinical practice will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 6 months to 11 years old at baseline.
* Patients with severe Atopic dermatitis (AD) according to the investigator's assessment.
* Patients initiating dupilumab (in those patients initiated retrospectively 2 months before the start of the study, the baseline information must be correctly filled out in the medical records).
* Signed informed consent by the parent/legally acceptable representative and assent by the patient appropriate to the patient's age.

Exclusion Criteria:

* Patients who are participating in an interventional clinical trial that modifies patient care.

Ages: 6 Months to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients aged 6 months to 11 years old at baseline and initiating Dupilumab for their Severe Atopic dermatitis (AD) in Spain.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-11-23 (Estimated)

PRIMARY OUTCOMES:
Demographic characteristic of pediatric patients initiating treatment with dupilumab for Severe AD: Age | At baseline
Demographic characteristic of pediatric patients initiating treatment with dupilumab for Severe AD: Gender | At baseline
Characteristic of pediatric patients initiating treatment with dupilumab for Severe AD:Body mass index (BMI) | At baseline
Medical history characteristics of pediatric patients initiating treatment with dupilumab for Severe AD | At baseline
  Including course of AD, recent AD treatment history, family history.
Medical history of atopic comorbidities | At baseline
  Selected atopic comorbidities over time will be reported.
Medical history of non-atopic diseases | At baseline

SECONDARY OUTCOMES:
Description of real-world treatment patterns: Dupilumab dosage | From baseline up to 24 months
Description of real-world treatment patterns: Dupilumab frequency of administration | From baseline up to 24 months
Description of real-world treatment patterns: Dupilumab reason for discontinuation | From baseline up to 24 months
  Reason for discontinuation will be reported if applicable.
Description of real-world treatment patterns (other treatments): Other type of treatment | From baseline up to 24 months
  In case of receiving other treatments for AD, topical or systemic.
Description of real-world treatment patterns (other treatments): Name of treatment | From baseline up to 24 months
  In case of receiving other treatments for AD, topical or systemic.
Description of real-world treatment patterns (other treatments): Duration of treatment | From baseline up to 24 months
  In case of receiving other treatments for AD, topical or systemic.
Description of real-world treatment patterns (other treatments): Reason for discontinuation (if applicable) | From baseline up to 24 months
  In case of receiving other treatments for AD, topical or systemic. Reason for discontinuation will be reported if applicable.
Participant-caregiver assessment: Change from baseline in the Children's Dermatology Life Quality Index score | From baseline up to 24 months
  The Children's Dermatology Life Quality Index (cDLQI) it is a 10-item questionnaire that assesses six different aspects that may affect quality of life, including symptoms and feelings, daily activities, leisure, work and school performance, personal relationships, and treatment. Each of the 10 questions is scored from 0 (not at all) to 3 (very much) and the overall cDLQI is calculated by summing the score of each question, resulting in a total score between 0-30. The higher the score, the more quality of life is impaired.
Participant-caregiver assessment: Change from baseline in the Infant's Dermatology Life Quality Index score | From baseline up to 24 months
  The Infant Dermatology Quality of Life Index (iDLQI) contains 10 questions and a response scale divided into four boxes. Each box gives a point between 0 and 3. The lower number is understood as the most positive for the participant.
  The index is filled out by a parent to a participating child between the ages of 0 to 5 years.
  Points from each question are added together and the end-sum represents the score. The sum score can be between 0 and 30. The higher the score the worse the assumed quality of life.
Participant-caregiver assessment: Change from baseline in the Dermatitis Family Impact (DFI) questionnaire | From baseline up to 24 months
  The DFI is a 10-item disease specific questionnaire assessing the impact of having a child with AD on family Quality of Life (QoL). The DFI questions are scored ranging from 0 to 3, and the total DFI score ranges from 0 to 30. The time frame of reference is the past week, and a higher DFI score indicates greater impairment in family QoL as affected by AD.
Participant-caregiver assessment: Change from baseline in the patient's Worst Itch Numerical Rating Scale (WI-NRS) | From baseline up to 24 months
  WI-NRS is a validated measure of itch severity. Patients will be asked daily to rate the intensity of their worst pruritus (itch) over the past 24 hours, using a 11-point scale ranging from 0 (no itch) to 10 (worst imaginable itch). Higher scores indicate more severity.
Caregiver assessment: Change from baseline in the patient's Worst Itch Scale Numerical Rating Scale (WSI-NRS) | From baseline up to 24 months
  The WSI-NRS is a single-item caregiver-reported. The caregivers describe their child "scratch" or "itch" in the AD-affected area by using numeric response options (0: no scratching/itching to 10: worst scratching/itching). Higher scores indicate more severity.
Physician assessment: Change from baseline in the eczema severity using the Eczema Area and Severity Index (EASI) | From baseline up to 24 months
  The EASI is calculated by summing 4 separate scores of the (1) head/neck, (2) upper extremities, (3) trunk, and (4) lower extremities. For each of the 4 anatomical regions, the score formula is SxAxM ["S" is the congregate score from the severity of 4 signs: erythema, oedema/papulation, excoriation, and lichenification graded on a discrete scale from 0 to 3, where 0 = absent, 1 = mild, 2 = moderate, and 3 = severe, giving S a maximum of 12. "A" represents the area to which AD affects the body, yielding a maximum of 6 points: 0 = 0%, 1 = 1-9%, 2 = 10-29%, 3 = 30-49%, 4 = 50-69%, 5 = 70-89%, and 6 = 90-100%. "M" is a multiplier, which is 0.1, 0.2, 0.3, and 0.4, respectively, for the region affected in those ≥8 years and 0.2, 0.2, 0.3, and 0.3, respectively, for those <8 years. The final EASI score is calculated based on the sum of the scores from the 4 anatomical regions. A higher score means higher AD severity. Scores range from 0 (no disease) to 72 (maximal disease severity).
Physician assessment: Percent change from beseline in the Body Surface Area (BSA) (%) affected by AD | From baseline up to 24 months
  BSA affected by AD disease will be assessed for each major section of the body (head, neck, anterior trunk, back, upper limbs, lower limbs, and genitals). It will be reported as a percentage of all major body sections combined.
Physician assessment: Change in Proportion of patients with Validated Investigator's Global Assessment (IGA) | From baseline up to 24 months
  The IGA is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
Physician assessment: Change from baseline in Biomarkers | From baseline up to 24 months
  Biomarker analysis will be performed, if available, in routine clinical practice and at routine visits
Number of Adverse Events (AE) / Serious Adverse Events (SAE) / Adverse Event of Special Interest (AESI) | From date of signed ICF, up to 24 months
  The number of events and the percentage of patients who had at least one event will be described.
Health Care Resource Utilization (HCRU) Questionnaire | From baseline up to 24 months
  Health care resource utilization may include hospitalizations (including length of stay), outpatient visits, urgent care or emergency room visits.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (15):
- Spain (15):
  - Investigational Site Number : 7240004, Santiago de Compostela, A Coruña [La Coruña]
  - Investigational Site Number : 7240006, Esplugues de Llobregat, Barcelona [Barcelona]
  - Investigational Site Number : 7240005, Oviedo, Principality of Asturias
  - Investigational Site Number : 7240008, Seville, Sevilla
  - Investigational Site Number : 7240002, Alicante
  - Investigational Site Number : 7240003, Barcelona
  - Investigational Site Number : 7240001, Madrid
  - Investigational Site Number : 7240010, Madrid
  - Investigational Site Number : 7240007, Madrid
  - Investigational Site Number : 7240014, Madrid
  - Investigational Site Number : 7240013, Málaga
  - Investigational Site Number : 7240012, Palma
  - Investigational Site Number : 7240009, San Cristóbal de La Laguna
  - Investigational Site Number : 7240016, Valencia
  - Investigational Site Number : 7240011, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org